CLINICAL TRIAL: NCT01266642
Title: Randomized Trial of Hypofractionated Whole Breast Irradiation Versus Conventionally Fractionated Whole Breast Irradiation for Ductal Carcinoma In Situ and Early Invasive Breast Cancer
Brief Title: Hypofractionated Radiation Therapy or Standard Radiation Therapy in Treating Patients With Ductal Breast Carcinoma In Situ or Early Invasive Breast Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2010-0559; NCI-2011-00253 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2010-0559 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2010-12-20; First posted 2010-12-24 (Estimated); Results first posted 2021-11-19 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Ductal Breast Carcinoma In Situ; Invasive Breast Carcinoma; Stage I Breast Cancer AJCC v6; Stage IA Breast Cancer AJCC v7; Stage IB Breast Cancer AJCC v7; Stage II Breast Cancer AJCC v6 and v7; Stage IIA Breast Cancer AJCC v6 and v7; Stage IIB Breast Cancer AJCC v6 and v7
MeSH Terms: conditions — Carcinoma, Intraductal, Noninfiltrating; Breast Neoplasms | interventions — Radiation; Radiation Dose Hypofractionation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I (HF-WBI) (Experimental): Patients undergo HF-WBI comprising external beam RT 5 days a week for approximately 3 weeks.
  Interventions: Radiation: External Beam Radiation Therapy; Radiation: Hypofractionated Radiation Therapy; Other: Laboratory Biomarker Analysis; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Radiation: Whole Breast Irradiation
- Arm II (CF-WBI) (Active Comparator): Patients undergo CF-WBI comprising external beam RT 5 days a week for approximately 5 weeks.
  Interventions: Radiation: External Beam Radiation Therapy; Other: Laboratory Biomarker Analysis; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Radiation: Whole Breast Irradiation

INTERVENTIONS:
Radiation: External Beam Radiation Therapy — Undergo HF-WBI
  Other Names: Definitive Radiation Therapy; EBRT; External Beam Radiation; External Beam Radiotherapy; External Beam RT; external radiation; External Radiation Therapy; external-beam radiation; Radiation, External Beam
  Arms: Arm I (HF-WBI)
Radiation: External Beam Radiation Therapy — Undergo CF-WBI
  Other Names: Definitive Radiation Therapy; EBRT; External Beam Radiation; External Beam Radiotherapy; External Beam RT; external radiation; External Radiation Therapy; external-beam radiation; Radiation, External Beam
  Arms: Arm II (CF-WBI)
Radiation: Hypofractionated Radiation Therapy — Undergo HF-WBI
  Other Names: Hypofractionated Radiotherapy; hypofractionation
  Arms: Arm I (HF-WBI)
Other: Laboratory Biomarker Analysis — Optional correlative studies
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies
Radiation: Whole Breast Irradiation — Undergo HF-WBI
  Arms: Arm I (HF-WBI)
Radiation: Whole Breast Irradiation — Undergo CF-WBI
  Arms: Arm II (CF-WBI)

SUMMARY:
This randomized phase II trial studies how well hypofractionated radiation therapy (RT) works compared to standard RT in treating patients with ductal breast carcinoma in situ (DCIS) or early invasive breast cancer. Radiation therapy (RT) uses high energy x-rays to kill tumor cells. Giving higher doses of RT over a shorter period of time may kill more tumor cells and have fewer side effects. It is not yet known if hypofractionated RT is more effective than standard RT in treating breast cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To compare patient-reported cosmetic outcome at 3 years using the Breast Cancer Treatment Outcomes Scale (BCTOS) for patients assigned to hypofractionated whole breast irradiation (HF-WBI) versus conventionally fractionated whole breast irradiation (CF-WBI).

SECONDARY OBJECTIVES:

I. To determine patient-reported cosmetic outcome using the BCTOS at 6 months, 1, 2, 4, and 5 years.

II. To determine physician-rated cosmetic outcome at 6 months, 1, 2, 3, 4, and 5 years using the Radiation Therapy and Oncology Group (RTOG) scale for physician assessment.

III. To determine the level of agreement between patient-rated cosmetic outcome and physician-rated cosmetic outcome at the various time points assessed.

IV. To determine the 5-year and risk of pathologically-confirmed invasive and/or in situ ipsilateral breast tumor recurrence (IBTR) for patients with ductal carcinoma in situ (DCIS) and early invasive breast cancer.

V. To determine patient-reported functional status and breast pain using the BCTOS at 6 months, 1, 2, 3, 4, and 5 years after treatment.

VI. To determine maximal acute (within 6 weeks of treatment) and late (more than 6 weeks after treatment) skin and soft tissue toxicities using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version (v)4.0 scale.

VII. To determine the relationship between the volume of breast tissue receiving excessive dose (defined as greater than 105% of the prescription dose) and the risk of adverse cosmesis.

VIII. To determine the relationship between bra cup size and the risk of adverse cosmesis.

IX. To determine whether there is a statistical interaction between breast volume and volume of tissue receiving greater than 105% of the prescription dose in predicting adverse cosmesis.

X. To determine in an exploratory analysis whether any other demographic, clinical, and pathologic factors correlate with risk of adverse cosmesis, quality of life, body image, image investment, and risk of IBTR.

XI. To determine if the C-509T variant allele of transforming growth factor-beta (TGF-beta) is associated with an increased risk of grade 2 or higher fibrosis (as determined by the Subjective, Objective, Medical Management, Analytic [SOMA] scale) three years after completion of radiation.

XII. To compare the cost of radiation for patients treated on the two treatment arms.

XIII. To compare patient quality of life, body image, and appearance investment for the two treatment arms using the Functional Assessment of Cancer Therapy-Breast (FACT-B), Appearance Schemas Inventory-Revised (ASI-R), and Body Image Scale, respectively.

XIV. To contribute additional blood samples to protocol LAB02-086 which is a case-control study investigating deoxyribonucleic acid (DNA) repair phenotypes and genotypes in breast cancer.

XV. To assess the psychometric profile of the Functional Assessment of Cancer Therapy-Breast (FACT-B) version 4 in collaboration with investigators from the Department of Medical Social Science, Northwestern University Feinberg School of Medicine.

XVI. To determine the influence of oncoplastic lumpectomy on the following outcomes: physician- and patient-reported cosmetic outcomes, other patient-reported health-related quality of life outcomes, and photographic measurements of breast cosmetic outcome.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients undergo HF-WBI comprising external beam RT 5 days a week for approximately 3 weeks.

ARM II: Patients undergo CF-WBI comprising external beam RT 5 days a week for approximately 5 weeks.

After completion of study treatment, patients are followed up at 6 months and then annually for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed ductal carcinoma in situ of the breast or early invasive breast cancer defined as pathologic stage Tis, T1, or T2, N0, N1mic, or N1a (pathologic staging of the axilla is required for all patients with invasive disease but is not required for patients with ductal carcinoma in situ [DCIS] only); (upfront pathologic stage cannot be assigned to patients treated with neoadjuvant chemotherapy; for such patients, the criteria for pathologic stage shall be applied to the initial clinical stage)
* Treatment with breast conserving surgery
* Final surgical margins must be negative, defined as no evidence for ductal carcinoma in situ or invasive breast cancer touching the inked surgical margin; if the invasive or in situ breast cancer approaches within less than 1 mm of the final surgical margin, then a re-excision is strongly encouraged; lobular carcinoma in situ at the final surgical margin will be disregarded
* Age 40 years or older. This age cutoff is justified because breast cancers in women under the age of 40 are known to have a significantly higher risk of IBTR presumably due to underlying biologic differences.
* Female sex.
* Attending radiation oncologist declares intention to treat the whole breast only and that a third radiation field to treat regional lymph nodes is not planned (radiation of the undissected level I/II axilla with high tangents is allowed)
* If the patient has a history of a prior non-breast cancer, all treatment for this cancer must have been completed prior to study registration and the patient must have no evidence of disease for this prior non-breast cancer
* Patients must be enrolled on the trial within 12 weeks of the later of two dates: the final breast conserving surgical procedure or administration of the last cycle of concurrent cytotoxic chemotherapy

Exclusion Criteria:

* Pathologic or clinical evidence for a stage T3 or T4 breast cancer
* Pathologic evidence for involvement of 4 or more axillary lymph nodes, or imaging evidence of involvement of infraclavicular, supraclavicular, or internal mammary lymph nodes
* Clinical or pathologic evidence for distant metastases
* Any prior diagnosis of invasive or ductal carcinoma in situ breast cancer in either breast
* Current diagnosis of bilateral breast cancer
* History of therapeutic irradiation to the breast, lower neck, mediastinum or other area in which there could potentially be overlap with the affected breast
* Patients not fluent in English or Spanish (The BCTOS will be available in these two languages)
* Patient is pregnant

Min Age: 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 301 (Actual)
Dates: Start 2011-02-08 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2025-11-30 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin D Smith, Principal Investigator — M.D. Anderson Cancer Center
Locations (7):
- United States (7):
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - UF Cancer Center at Orlando Health, Orlando, Florida
  - MD Anderson in The Woodlands, Conroe, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - MD Anderson West Houston, Houston, Texas
  - MD Anderson League City, League City, Texas
  - MD Anderson in Sugar Land, Sugar Land, Texas

REFERENCES:
- [Derived] Weng JK, Lei X, Schlembach P, Bloom ES, Shaitelman SF, Arzu IY, Chronowski G, Dvorak T, Grade E, Hoffman K, Perkins G, Reed VK, Shah SJ, Stauder MC, Strom EA, Tereffe W, Woodward WA, Hortobagyi GN, Hunt KK, Buchholz TA, Smith BD. Five-Year Longitudinal Analysis of Patient-Reported Outcomes and Cosmesis in a Randomized Trial of Conventionally Fractionated Versus Hypofractionated Whole-Breast Irradiation. Int J Radiat Oncol Biol Phys. 2021 Oct 1;111(2):360-370. doi: 10.1016/j.ijrobp.2021.05.004. Epub 2021 May 13. PMID 33992718
- [Derived] Grossberg AJ, Lei X, Xu T, Shaitelman SF, Hoffman KE, Bloom ES, Stauder MC, Tereffe W, Schlembach PJ, Woodward WA, Buchholz TA, Smith BD. Association of Transforming Growth Factor beta Polymorphism C-509T With Radiation-Induced Fibrosis Among Patients With Early-Stage Breast Cancer: A Secondary Analysis of a Randomized Clinical Trial. JAMA Oncol. 2018 Dec 1;4(12):1751-1757. doi: 10.1001/jamaoncol.2018.2583. PMID 30027292
- [Derived] Shaitelman SF, Schlembach PJ, Arzu I, Ballo M, Bloom ES, Buchholz D, Chronowski GM, Dvorak T, Grade E, Hoffman KE, Kelly P, Ludwig M, Perkins GH, Reed V, Shah S, Stauder MC, Strom EA, Tereffe W, Woodward WA, Ensor J, Baumann D, Thompson AM, Amaya D, Davis T, Guerra W, Hamblin L, Hortobagyi G, Hunt KK, Buchholz TA, Smith BD. Acute and Short-term Toxic Effects of Conventionally Fractionated vs Hypofractionated Whole-Breast Irradiation: A Randomized Clinical Trial. JAMA Oncol. 2015 Oct;1(7):931-41. doi: 10.1001/jamaoncol.2015.2666. PMID 26247543
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from provider clinics at 3 academic medical centers between February 2011 and February 2014. Women with stage 0 to II breast cancer were randomly assigned to CF-WBI or HF-WBI, stratified by chemotherapy, margin status, cosmesis, and breast size.
Pre-assignment Details: Of the 301 participants enrolled, 287 were fully eligible and were randomized to protocol, 13 were excluded (8) Insurance would not cover protocol therapy, (4) withdrew consent and (1) became ineligible due to finding of other primary cancer on simulation CT. 1 participant was registered twice.
Groups:
- CF-WBI: 50 Gy in 25 fractions to the whole breast, plus a tumor bed boost of 10Gy in 5 fractions or of 14Gy in 7 fractions (dependent on surgical margins).
- HF-WBI: 42.56 Gy in 16 fractions to the whole breast, plus tumor bed boost of 10Gy in 4 fractions or 12.5Gy in 5 fractions (dependent on surgical margins).
Period: Overall Study
Arm/Group | CF-WBI | HF-WBI
Started | 149 | 138
Completed | 149 | 137
Not Completed | 0 | 1
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CF-WBI | HF-WBI | Total
Number analyzed (Participants) | 149 | 138 | 287
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.3 (8) | 60 (8.6) | 60.2 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 149 | 138 | 287
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 16 | 20 | 36
  Not Hispanic or Latino | 133 | 118 | 251
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 17 | 17 | 34
  White | 130 | 119 | 249
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 149 | 138 | 287

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Scores of Either <2.5 or >=2.5 on the Breast Cancer Treatment Outcome Scale (BCTOS) Cosmesis
Description: BCTOS cosmesis score range from 1 to 4, and scores of 2.5 or more indicate adverse cosmetic outcomes.
Time Frame: 3 years after completing radiation therapy
Population: Intent to treat population (all participants assigned to CF-WBI or HF-WBI).
Measure: Count of Participants; unit: Participants
Arm/Group | CF-WBI | HF-WBI
Number analyzed (Participants) | 149 | 138
Participants
  BCTOS cosmesis < 2.5 | 97 | 88
  BCTOS cosmesis >= 2.5 | 17 | 15
  Unknown | 35 | 35

2. Secondary Outcome: Panel Physicians Rated Cosmesis
Description: A group of three attending physicians blinded to the treatment scored the photographs using the Radiation Therapy and Oncology Group (RTOG) criteria. RTOG scale range from 1 (excellent), 2 (good), 3 (fair), and 4 (poor).
Time Frame: 3 years after completing radiation therapy.
Population: Intent to treat population (all participants assigned to CF-WBI or HF-WBI).
Measure: Count of Participants; unit: Participants
Arm/Group | CF-WBI | HF-WBI
Number analyzed (Participants) | 149 | 138
Participants
  Excellent/Good | 86 | 72
  Fair/Poor | 28 | 31
  Unknown | 35 | 35

ADVERSE EVENTS:
Time Frame: From the time radiotherapy was completed until 5-years post treatment.
Arm/Group | CF-WBI | HF-WBI
All-Cause Mortality (participants affected / at risk) | 0/149 | 1/138
Serious Adverse Events (participants affected / at risk) | 0/149 | 0/138
Other Adverse Events (participants affected / at risk) | 149/149 | 138/138
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CF-WBI (N=149) | HF-WBI (N=138)
Fatigue (General disorders) | 135 | 114
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 132 | 109
Skin induration (Skin and subcutaneous tissue disorders) | 39 | 45
Dermatitis (Skin and subcutaneous tissue disorders) | 148 | 130
Telangiectasia (Skin and subcutaneous tissue disorders) | 17 | 18
Lymphedema (Vascular disorders) | 12 | 7
Superficial soft tissue fibrosis (Musculoskeletal and connective tissue disorders) | 89 | 79
Fibrosis deep connective tissue (Musculoskeletal and connective tissue disorders) | 50 | 51
Seroma (Injury, poisoning and procedural complications) | 36 | 40
Breast pain (Reproductive system and breast disorders) | 123 | 100
Cough (Respiratory, thoracic and mediastinal disorders) | 9 | 9
Nipple deformity (Respiratory, thoracic and mediastinal disorders) | 61 | 49
Breast atrophy (Reproductive system and breast disorders) | 105 | 96
Pruritus (Skin and subcutaneous tissue disorders) | 120 | 75

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-08-16): https://cdn.clinicaltrials.gov/large-docs/42/NCT01266642/Prot_SAP_000.pdf